CLINICAL TRIAL: NCT01113905
Title: Beta-Endorphin as a Mediator of Cancer Therapy-Induced Fatigue
Brief Title: Role of Beta-Endorphin in Cancer Therapy Fatigue
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment was obtained
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David E. Fisher, M.D., Ph.D, Chairman, Dept of Dermatology, Massachusetts General Hospital
Other Study IDs: 09-222
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer; Fatigue
Keywords: Fatigue; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to be measured for levels of beta-endorphin
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Radiation Only
- Radiation and Chemotherapy

SUMMARY:
The investigators aim to test whether beta-endorphin, a substance our bodies make in response to painful and stressful stimuli, plays a causative role in radiation-induced fatigue that cancer patients receiving radiation therapy commonly experience. If this is so, the investigators' hope is to direct efforts at treating radiation-induced fatigue using agents that block the action of beta-endorphin with the aim of improving quality of life for patients undergoing radiation therapy

DETAILED DESCRIPTION:
Participants will be breast cancer patients receiving radiation therapy at Massachusetts General Hospital. There will be two groups of patients: those receiving adjuvant radiation therapy alone following surgical tumor resection, and those receiving adjuvant chemotherapy and radiation therapy following surgical tumor resection. Patients receiving any radiation regimen detailed below in section 2b are eligible for the study. In this study the investigators will be drawing blood for beta-endorphin measurement prior to, at various times during, and following patients' treatment regimens. In addition, at each blood draw, patients will complete questionnaires that assess fatigue, mood, and pain. These questionnaires have all been validated for use in cancer patients (see "Procedures Involving Human Participants section below), and for our study, the investigators have formatted them onto computer tablets for ease of patient completion and data analysis. This study will progress as follows:

Patients: Patients expected to receive adjuvant radiation therapy at Massachusetts General Hospital will be approached for enrollment onto this study. Two groups of patients, a chemotherapy group and a non-chemotherapy group, will be enrolled as follows:

1. Adjuvant chemotherapy followed by radiation therapy
2. Adjuvant radiation therapy without chemotherapy

The enrollment goal for each group is 50 patients (total of 100 patients for the study). This calculation is based on the approximate number of 30 patients the investigators will need to achieve a sensitivity of β-endorphin changes of 5 pM being statistically significant to a p-value of<0.05 with 95% power. Based in our finding in mice, the investigators expect β-endorphin levels to vary between individuals, and the investigators have increased sample size by 70% from our calculations to account for deviations from our β-endorphin levels estimations. Additionally, the investigators have added patients to account for a number of patient dropping out of the study, since this is a long trial for patients requiring multiple blood draws.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Pathologic diagnosis of stage 0-III breast cancer (any histologic subtype) in either breast or both breasts
3. Previous resection of tumor, either by mastectomy or partial mastectomy, ±sentinel lymph node biopsy, ±axillary lymph node dissection
4. A likelihood of having radiation therapy or chemotherapy following surgery as determined by the on-site principal investigator (PI) or co-investigator
5. Signed informed consent which has been reviewed and approved by the Institutional Review Board and no condition that impairs the ability to provide informed consent (e.g. uncontrolled psychiatric illness)

Eligibility for the radiation therapy (RT) alone group will include:

1. Planned 3-D conformal radiation therapy to the whole breast (2 tangential fields, unilateral or bilateral) via standard or Canadian Fractionation, +/- regional nodal irradiation.
2. No planned chemotherapy for this tumor

Eligibility for the RT + chemotherapy (CT) group will include:

1. Planned 3-D conformal radiation therapy to the whole breast (2 tangential fields, unilateral or bilateral) via standard or Canadian fractionation (photons followed by a photon, electron, or mixed photon/electron boost), +/- regional nodal irradiation.
2. Planned adjuvant chemotherapy (any regimen except for biologic therapy alone)

Exclusion Criteria:

1. Continuous/chronic treatment with opiate/opioid analgesics for 3-6 months prior to enrollment. In addition, patients receiving radiation therapy alone who have taken opiate analgesics from their surgery within 72 hours of the post-surgery/pre-radiation therapy blood draw (at 1-6 weeks prior to the start of radiation therapy) will be removed from the study. Patients receiving chemotherapy and radiation therapy who have taken opiate analgesics from their surgery within 72 hours of the blood draw prior to cycle 1 of chemotherapy will be removed from the study.
2. Prior radiation therapy to the chest or brain
3. Patients diagnosed with Stage IV breast cancer
4. History of illegal drug use within 6 months prior to enrollment
5. At point of enrollment, diagnosis of major depression, bipolar disorder, seasonal affective disorder, or anxiety disorder for which the patient is currently taking any of the following medications: selective serotonin reuptake inhibitors (SSRIs), Tricyclic antidepressants, monoamine oxidase inhibitors, lithium, benzodiazepines, barbiturates, drugs acting on the 5-HT receptors. Patients meeting these criteria may still enroll in the study if they are on a chronic, stable, low-dose regimen for at least 3 months prior to enrollment, as determined by the on-site PIs and co-investigating physicians. Patients having to begin on a regimen of any of these medications while on the study may continue on the study.
6. Anemia of any etiology at initial visit (Hct <33%) and the following baseline fatigue scores on the Fatigue Symptom Inventory (FSI): Average score for question #s 1-4 > 5; and/or Average score for question #s 5-11 > 5. Patients with Hct<33% but who have no baseline fatigue (as indicated by baseline scores on the FSI as follows: average score for question #s 1-4 < 5 and average scores for question #s 5-11 < 5) are eligible to participate.
7. Endocrine disorders that can cause fatigue: Addison's disease, uncorrected hypothyroidism (patients taking thyroid replacement therapy for at least 3 months prior to enrollment patients are eligible), central endocrine deficiency, polyglandular autoimmune failure.
8. Patients with thyroid disease (hypothyroidism or hyperthyroidism) that was diagnosed within 3 months of cancer diagnosis or patients with previously stable thyroid disease who have experienced symptoms or have had to change their medication doses within 3 months of cancer diagnosis. Patients with stable disease who have no had to change medication doses within 3 months of cancer diagnosis. Patients with stable disease who have not had to change medication doses within 3 months of cancer diagnosis may enroll as long as baseline fatigue scores do not meet criteria for exclusion. Patients enrolled in the study who have to alter doses of thyroid medications or who are newly diagnosed with thyroid disease while on the study will be removed from the study, and will not count towards our total patient accrual.
9. Uncontrolled autoimmune diseases that can cause fatigue, including fibromyalgia and fatigue syndromes. If these are controlled, enrollment or maintenance of the patient on the protocol may continue at the discretion of the enrolling principal investigator.
10. Sleep disorder diagnosed within 3 months of enrollment and the following baseline fatigue scores on the FSI: Average score for question #s 1-4 > 5; and/or average score for question #s 5-11 > 5. Patients diagnosed with a sleep disorder within 3 months of enrollment and with FSI scores < 5 on question #s 1-4 and #s 5-11 are eligible.
11. Activity-limiting heart or lung disease
12. Renal failure (BUN and creatinine should be within the normal range for the prior 6 months)
13. Baseline fatigue as indicated by the following baseline scores on the FSI: Average score for question #s 1-4 > 5; and/or Average score for question #s 5-11 > 5.
14. Patients receiving chemotherapy or radiation therapy at any site other than Massachusetts General Hospital
15. Hepatitis or chronic liver disease (albumin <3 g/dL or >6 g/dL; ALT >60 U/L or < 5 U/L, AST > 40 U/L or <5 U/L)
16. Untreated chronic infection (e.g. tuberculosis, osteomyelitis, abscess). Patients being treated for these may be enrolled in, or continue on the protocol at the discretion of the principal investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who plan to have radiation therapy only or radiation therapy and chemotherapy after their mastectomy or lumpectomy.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
correlation of endorphin level to fatigue questionnaire results | one year

CONTACTS AND LOCATIONS:
Overall Officials: David E Fisher, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States